CLINICAL TRIAL: NCT07037004
Title: Impact of Microbiome Modulation With CBM588 in Combination With Pembrolizumab for Adjuvant Therapy of High-Risk, Resected Renal Cell Carcinoma (RCC)
Brief Title: Adding a Live Biotherapeutic Product (CBM588) to Pembrolizumab for the Treatment of Renal Cell Cancer After Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24709; NCI-2025-04100 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24709 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-06-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Clear Cell Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage II Renal Cell Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (CBM588, pembrolizumab) (Experimental): Patients receive CBM588 PO BID on days 1-21 or days 1-42 of each cycle and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Clostridium butyricum CBM588 Strain; Procedure: Computed Tomography; Biological: Pembrolizumab
- Arm 2 (pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Clostridium butyricum CBM588 Strain — Given PO
  Other Names: C. butyricum CBM588 Strain; C. butyricum MIYAIRI Strain; C. butyricum Strain MIYAIRI 588; CBM588; Clostridium butyricum MIYAIRI 588; Clostridium butyricum MIYAIRI 588 Strain; MIYAIRI 588; MIYAIRI 588 Strain of C. butyricum
  Arms: Arm 1 (CBM588, pembrolizumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase II trial compares the effect of adding a Live Biotherapeutic Product called CBM588 to pembrolizumab versus pembrolizumab alone in preventing return of disease (recurrence) after surgery for patients with renal cell cancer. Pembrolizumab is an immune checkpoint inhibitor. Immunotherapy with monoclonal antibodies such as pembrolizumab may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pembrolizumab is approved for the treatment of renal cell cancer after surgery. Research has shown that changes to the composition of the healthy bacteria in the body (the microbiome), may improve a patient's response to treatment with immunotherapy. CBM588, a Live Biotherapeutic Product (LBP) containing a bacteria called Clostridium butyricum, has been shown to improve outcomes in patients treated with immunotherapy for other types of cancer. Adding CBM588 to treatment with pembrolizumab after surgery may cause changes in the microbiome that improve patient response to treatment and reduce disease recurrence, compared to pembrolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the Clostridium butyricum CBM588 strain (CBM588) increases interleukin (IL)-12 production in patients with high-risk, resected renal cell carcinoma (RCC) receiving pembrolizumab.

SECONDARY OBJECTIVES:

I. To determine if CBM588 improves recurrence-free survival (RFS) in patients with high-risk, resected renal cell carcinoma (RCC) receiving pembrolizumab.

II. To determine if CBM588 improves overall survival (OS) in patients with high-risk, resected renal cell carcinoma (RCC) receiving pembrolizumab.

III. To characterize global changes in stool microbiome profile in patients with high-risk, resected RCC receiving pembrolizumab with or without CBM588.

IV. To characterize changes in circulating cytokine and immune cell populations in patients with high-risk, resected RCC receiving pembrolizumab with or without CBM588.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive CBM588 orally (PO) twice daily (BID) on days 1-21 or days 1-42 of each cycle and pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and computed tomography (CT) throughout the study.

ARM 2: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples and CT throughout the study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide informed consent for the trial
* Histological confirmation of renal cell carcinoma (RCC) with a clear-cell or sarcomatoid component
* Pathologic stage of pT2, G4 or sarcomatoid, N0M0; pT3, any grade, N0M0; pT4, any grade, N0M0; pTany, any grade, N+M0; or M1 no evidence of disease (NED) after resection
* No prior systemic immunotherapy for RCC
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Males and females, ages ≥ 18
* Any ethnicity or race
* Calculated creatinine clearance ≥ 30 milliliters per minute (mL/min) per the Cockcroft and Gault formula or serum creatinine < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN if liver metastases are present)
* Total bilirubin < 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin up to 3.0 mg/dL)
* Adequate bone marrow function defined by any of the following laboratory test findings: white blood cells (WBC) > 2,000/mm^3, neutrophils > 1,500/mm^3, platelets > 100,000/mm^3
* Female subjects of child-bearing potential and female partners of male subjects must agree to use a highly effective method of contraception during treatment and for at least 5 months after the last dose

  * Highly effective methods of contraception include: tubal ligation, an approved hormonal contraceptive such as oral contraceptives, patches, implants, injections, rings or hormonally impregnated intrauterine device (IUD), or IUD

Exclusion Criteria:

* Prior radiation or anti-PD1, anti-PDL1, or anti-CTLA-4 therapy for RCC
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids
* Baseline pulse oximetry less than 92% "on room air"
* Current use, or intent to use probiotics, prebiotics, yogurt, bacterial fortified foods and other natural supplements ≤ 2 weeks prior to treatment initiation and during the period of treatment
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Uncontrolled adrenal insufficiency
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Not recovered to ≤ grade 1 toxicities related to any prior therapy before administration of study drug
* Women who are pregnant or breastfeeding
* History of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), as well as unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-05-04 (Estimated); Primary Completion 2027-05-04 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Change in interleukin (IL)-12 levels | Baseline to week 12
  A two-sample t-test will be used to test the difference in the changes in IL-12 production for the two treatment arms. A Wilcoxon rank-sum test will be used if the changes are not normally distributed (p< 0.05 by a Shapiro-Wilks test).

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | From randomization to disease recurrence or death, assessed up to 1 year
  RFS will be estimated by the Kaplan-Meier method. Median RFS and landmark RFS rates (e.g., 1-year and 2-year RFS) will be calculated with confidence intervals. Log-rank test will be used to compare the distribution between groups. Cox proportional hazards model will be used to estimate hazard ratios with 95% confidence intervals.
Overall survival (OS) | From randomization to death from any cause, assessed up to 1 year
  OS will be estimated by the Kaplan-Meier method. Median OS and landmark OS rates (e.g., 1-year and 2-year OS) will be calculated with confidence intervals. Log-rank test will be used to compare the distribution between groups. Cox proportional hazards model will be used to estimate hazard ratios with 95% confidence intervals.
Shannon diversity index | Baseline to week 12
  A comparison of the Shannon diversity index (a measure of microbial diversity) from baseline to week 12 will be conducted.
Proportion of circulating regulatory T cells (Tregs) | Baseline to week 12
  Will estimate the proportion of Tregs in the blood.
Proportion of circulating myeloid derived suppressor cells (MDSCs) | Baseline to week 12
  Will estimate the proportion of MDSCs in the blood.
IL-6, IL-8 and other cytokines/chemokines | Baseline to week 12
  Will compare IL-6, IL-8 and other cytokines/chemokines.
Incidence of toxicities | Up to 30 days after last dose
  Toxicities such as diarrhea and nausea will be assessed using Common Terminology Criteria for Adverse Events version 5 criteria. Will perform statistical analysis to compare the rates of all grade and grade ≥ 3 treatment related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Yip, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California